CLINICAL TRIAL: NCT03217942
Title: Spread of Muscle Hyperalgesia and Pain in a Low Dose NGF-induced Pain Model
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Line Bay Sørensen, Ph.d. stud., Aalborg University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: N-2017-0007
Record Dates: First submitted 2017-07-10; First posted 2017-07-14 (Actual); Last update posted 2018-01-11 (Actual); Status verified 2018-01

CONDITIONS: Hyperalgesia; Healthy Subjects
Keywords: Muscle soreness; NGF-induced pain; Pain model; Long-lasting sensitization
MeSH Terms: conditions — Hyperalgesia; Myalgia | interventions — Nerve Growth Factor

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low dose (Experimental): All participants will receive 5 i.m injections of NGF (1 ug/0.5ml) into the tibialis anterior muscle (either left or right leg)
  Interventions: Drug: NGF
- High dose (Experimental): All participants will receive 1 high dose i.m bolus injection of NGF (5 ug/0.5ml) and 4 injections of saline (control/same volume) into the tibialis anterior muscle (either left or right leg)
  Interventions: Drug: NGF

INTERVENTIONS:
Drug: NGF — Intramuscular injection
  Other Names: Beta-Nerve Growth Factor, Human

SUMMARY:
The purpose of this study is to investigate and determine the time course and distribution on muscle hyperalgesia and muscle pain in a repeated, low dose NGF model. It is hypothesized that low dosages i.m injections of NGF are able to induce mechanical hyperalgesia and muscle soreness in a same manner (effect of duration) as for dosages previously used in NGF studies. Furthermore, it is also speculated if several injections of low dose NGF into the muscle combined are able to course immediate pain sensation and spreading of muscle hypersensitivity.

DETAILED DESCRIPTION:
Effects of pain responses, symptom development and pattern (time course and distribution) following 5 i.m low dose injections of NGF injected into the tibialis anterior muscle will be compared to a high dose i.m injection of NGF injected into the contralateral side in healthy pain-free subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy and pain free volunteers

Exclusion Criteria:

* Pregnancy
* Drug addiction defined as the use of cannabis, opioids or other drugs
* Previous neurologic, mental illnesses, or psychiatric diseases.
* Past history of chronic pain in the musculoskeletal system (muscle, joint, cartilage, connective tissue)
* Participation in other pain trials throughout the study period
* Lack of ability to cooperate
* Taking any analgesic 24 hours before the injections
* Performing any strenuous leg exercise through out the study period causing sore muscles

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Muscle sensitivity | Change from baseline at 3 weeks
  Pressure pain thresholds (PPTs) are assessed over the tibialis anterior muscles using a handhold pressure algometer.

SECONDARY OUTCOMES:
Pressure-induced referred pain | Change from baseline at 3 weeks
  At three predetermined sites within the tibialis anterior muscle, a constant pressure stimulation (120% of PPT) is evoked by use of the pressure algometer. Subjects color their perceived sensation of pain on an electronic schematic of the lower legs using Navigate Pain.
Activity-induced muscle soreness | Change from baseline at 3 weeks
  Subjects perform 10 dorsiflexions with each leg. The perceived muscle soreness is reported using a numeric rating scale (NRS) and the area of soreness is colored on an electronic schematic of the lower legs (Navigate Pain).
Pain intensity | Assessed continuously at 0-5 min during the injections at each leg
  Subjects rate their perceived pain intensity on a visual analogue scale (VAS) App (Aalborg University) as displayed on a tablet computer with a sample rate of 1 Hz.
Muscle soreness Diary | Change from baseline at 3 weeks
  Two times a day subjects evaluate their muscle soreness using a Likert Scale of muscle soreness for lower limp
Activity-induced muscle soreness Diary | Change from baseline at 1 week
  Subjects perform 10 dorsiflexions with each leg. The perceived muscle soreness is reported using a numeric rating scale (NRS) and the area of soreness is colored on an electronic schematic of the lower legs (Navigate Pain). The activity is performed at home on days in between the sessions

CONTACTS AND LOCATIONS:
Overall Officials: Line Bay Sørensen, Ph.d stud., Principal Investigator — Aalborg University
Locations (1):
- Aalborg University, Aalborg, Denmark